CLINICAL TRIAL: NCT00158834
Title: Comparison of Stepwise Treatment of Asthmatic Children With Salmeterol/Fluticasone Propionate Combination Product (Seretide®) and/or Fluticasone Propionate (Flixotide®) Based on PD20 Methacholine and Symptoms or Based on Symptoms Only (Children Asthma Therapy Optimal)
Brief Title: Pediatric Asthma Study Using Stepwise Treatment With Two Food And Drug Administration Approved Asthma Medications
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAS30018; SER9702/CATO
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Asthma
Keywords: Children; Asthma; bronchial hyperresponsiveness; symptoms
MeSH Terms: conditions — Asthma; Bronchial Hyperreactivity | interventions — Salmeterol Xinafoate; Fluticasone

INTERVENTIONS:
Drug: Salmeterol/Fluticasone propionate combination product
Drug: Fluticasone propionate
  Other Names: Salmeterol/Fluticasone propionate combination product

SUMMARY:
This study was designed to evaluate if, in children with asthma, a stepwise treatment (five levels varying from once daily fluticasone propionate 100mcg until twice daily a fixed combination of salmeterol and fluticasone propionate 50/500 mcg) based on symptom scores alone results in a sub-optimal treatment when compared to treatment based on cumulative symptom scores and bronchial hyperresponsiveness (PD20 methacholine).

ELIGIBILITY:
Inclusion criteria:

* Children with a documented history of asthma.
* Using inhaled steroids from 100 mcg up to 500 mcg twice daily for at least 1 month before study start.
* Must be able to perform reproducible lung function tests.
* Must have a positive RAST or skin prick test.
* During the treatment period, the patient has to be hyperreactive (defined as PD20 methacholine < 150 mcg) and/or have a cumulative symptom score of 14 based on the daily record card filled in during the last 2 weeks of the run-in period.

Exclusion criteria:

* History of an acute upper or lower respiratory tract infection, middle ear, or sinus infection 4 weeks prior to visit 1.
* Admitted to hospital due to a respiratory disease 4 weeks prior to visit 1.
* Received oral corticosteroids within 4 weeks prior to visit 1.
* Existence of any disorder that affects growth.
* Clinical or laboratory evidence of a serious systemic disease, or suspected hypersensitivity to corticosteroids, lactose or short/long acting B2-agonists.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Start 1999-11

PRIMARY OUTCOMES:
Asthma symptom free days during the last 12 weeks of the treatment period.

SECONDARY OUTCOMES:
Bronchial hyperresponsiveness, determined by PD20 methacholine at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (15):
- Netherlands (15):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Hilversum
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sittard
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Veldhoven
  - GSK Investigational Site, Zwolle